CLINICAL TRIAL: NCT06863740
Title: Using Cannabis to Treat Restless Legs Syndrome: A Randomized Placebo Controlled Pilot Safety and Feasibility Trial
Brief Title: Using Cannabis to Treat Restless Legs Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4752
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Restless Leg Syndrome (RLS)
MeSH Terms: conditions — Restless Legs Syndrome | interventions — nabiximols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cannabis Arm (Experimental): 5:1 CBD:THC oral cannabis
  Interventions: Drug: Cannabis oil
- Placebo Arm (Placebo Comparator): Oral placebo
  Interventions: Drug: Cannabis placebo

INTERVENTIONS:
Drug: Cannabis oil — 5:1 CBD:THC oral formulation with a concentration of 25 mg/g CBD and 5 mg/g THC in a pharmaceutical grade medium chain triglyceride (MCT) oil.
  Other Names: MPL-005
  Arms: Cannabis Arm
Drug: Cannabis placebo — Placebo oil
  Arms: Placebo Arm

SUMMARY:
Restless Legs Syndrome (RLS) is a disorder that causes painful and uncomfortable sensations in the legs, and its symptoms have a significant impact on sleep and quality of life. Cannabis has been used by some RLS patients as a treatment due to its painkilling and drowsiness effects, however there has never been a clinical research trial investigating cannabis in patients with RLS. A controlled trial is needed to establish how safe and feasible cannabis is as a treatment for RLS. The investigators plan to randomize 30 participants with moderate-to-severe RLS to receive either cannabis or placebo for 8 weeks. The investigators will measure patients sleep quality and quality of life at baseline and 8-week follow-up. The investigators will also monitor patients for any adverse reactions to the study drug.

ELIGIBILITY:
Inclusion Criteria:

* ≥25 years of age
* diagnosis of RLS based on the International RLS Study Group criteria
* refractory RLS symptoms despite use of dopaminergic and/or alpha-2-delta ligand therapy
* onset of RLS at least 6 months before screening

Exclusion Criteria:

* sleep disordered breathing, or sleep disordered breathing that is not adequately controlled on therapy (apnea-hypopnea index of >15)
* cannabis use within 4 weeks of study enrollment
* known allergy to cannabis, cannabinoids or palm/coconut oil
* Currently pregnant or breast-feeding (a negative urine pregnancy test must be obtained for women of childbearing potential during pretreatment evaluation)
* Active substance abuse
* Ischemic heart disease with unstable angina or recent acute coronary syndrome in the last 3 months, uncontrolled arrhythmias, poorly controlled hypertension
* Serious liver disease
* History of schizophrenia or any other psychotic disorder

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events and Serious Adverse Events | 8 weeks
  We will measure the rate and type of treatment related adverse events
Rate of Study Completion | 8 weeks
  The percentage of enrolled participants who complete the study

SECONDARY OUTCOMES:
Change from Baseline in Restless Legs Syndrome Quality of Life (RLSQoL) at 8 Weeks | 8 weeks
  The Summary Score of the RLSQoL will be calculated, ranging from 0 (worse quality of life) to 100 (best quality of life).
Change from Baseline in Self-Reported Quality of Life on the Short Form-36 (SF-36) Health Survey Questionnaire at 8 Weeks | 8 weeks
  The SF-36 Questionnaire has 36-items that covers eight areas: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. Scores for each domain range from 0 to 100, with a higher score indicating better health.
Change in Restless Legs Syndrome Severity using the International RLS Study Group Rating Scale from Baseline to Follow-up | 8 weeks
  The International RLS Study Group Rating Scale measures RLS severity based on the following summary scale:
  Very severe=31-40 points Severe=21-30 points Moderate=11-20 points Mild=1-10 points None=0 points
Change in Sleep Quality as assessed by the Pittsburgh Sleep Quality Index from Baseline to Follow-Up | 8 weeks
  Sleep quality as assessed by the Pittsburgh Sleep Quality Index. The questionnaire is scored on a range from 0-21 points, with "0" indicating no difficulty and "21" indicating severe difficulties in all areas.
Change in Daytime Sleepiness as assessed by the Epworth Sleepiness Scale from Baseline to Follow-Up | 8 weeks
  Scores on Epworth Sleepiness Scale range from range from 0 to 24, with higher scores indicating higher average sleep propensity in daily life (daytime sleepiness).
Change in Mood as assessed by the Beck Depression Inventory from Baseline to Follow-Up | 8 weeks
  The Beck Depression Inventory has 21 questions that are scored on a range of 0-63 points. Higher scores indicate more severe depression.
Change in Objective Sleep Quality as Measured by Actigraphy from Baseline to Follow-Up | 8 weeks
  Objective sleep quality will be assessed using wrist actigraphy that will be provided with the home sleep apnea test. Sleep efficiency will be calculated by dividing the amount of time spent asleep (in minutes) by the total amount of time in bed (in minutes).
Change in Leg Movements as Measured by Ankle Actigraphy from Baseline to Follow-Up | 8 weeks
  Ankle actigraphy will be used to count the number of leg movements that occur throughout the night.
Change in Obstructive Sleep Apnea (OSA) Severity (as measured by the apnea-hypopnea index) from Baseline to Follow-Up | 8 weeks
  Measured by the apnea-hypopnea index (AHI). AHI quantifies the number of apneas and hypopneas per hour of sleep. It will be measured using a home sleep monitor or a readout from a continuous positive airway pressure (CPAP) machine.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No